CLINICAL TRIAL: NCT01724710
Title: To Study the Effect of Organic Light Emitting Diodes (OLED) on Cultured Fibroblast
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201206038RIC
Record Dates: First submitted 2012-08-28; First posted 2012-11-12 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Non-pressure Chronic Ulcer of Skin, Not Elsewhere Classified

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fibroblasts of Chronic ulcer and normal skin will be cultured. Fibroblast culture will be analyzed with quantitative PCR.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- chronic ulcer: 1x1cm2 tissue from chronic ulcer wound
- normal skin: 1x1x0.1 cm3 normal skin from graft

SUMMARY:
Chronic ulcers is a common clinical problem. Diabetes or peripheral vascular occlusion is major reason leading to chronic wound healing.

The investigators's previous animal experiments have confirmed that OLED can promote burn wound healing and fibroblast proliferation in normal Wistar rat.

In order to find the time point and dosage of the effective light therapy. The investigators further use cultured human fibroblasts in vitro to study light therapy to promote fibroblast proliferation mechanisms.

Expect clinical application of light therapy in the future is more accurate and effective.

DETAILED DESCRIPTION:
Chronic ulcers is a common clinical problem. Diabetes or peripheral vascular occlusion is major reason leading to chronic wound healing.

Therapeutic methods to promote wound healing are hyperbaric oxygen therapy, vacuum assisted therapy and photostimulation.

Although there are many treatments but no one has been widely accepted. The clinical effects of uncertainty, high cost and inconvenience of use is the main reason.

Each year amputation of the population due to chronic ulcers has not decreased. In order to break the current medical difficulties, We refer to the new light therapy technology.

Look forward to shorten the healing time and reduce medicine costs. The investigators's previous animal experiments have confirmed that OLED can promote burn wound healing and fibroblast proliferation in normal Wistar rat.

In order to find the time point and dosage of the effective light therapy. The investigators further use cultured human fibroblasts in vitro to study light therapy to promote fibroblast proliferation mechanisms.

Expect clinical application of light therapy in the future is more accurate and effective irradiative time points and dosage.

ELIGIBILITY:
Inclusion Criteria:

* chronic ulcer
* normal skin
* age 50~80 years,
* chronic skin ulcer patient
* skin-grafting patient

Exclusion Criteria:

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. The process of collecting chronic ulcer skin: When the patient accept wound debridement surgery, visiting staff will take 1x1cm2 skin of chronic ulcer.
  2. The process of collecting normal skin: When the patient accept skin-grafting surgery, visiting staff will take 1x1x0.1cm3 skin.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kean Eng Yeong, college, Study Chair — NTUH Burn lab
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan